CLINICAL TRIAL: NCT00001384
Title: A Pilot Trial of AC (Adriamycin, Cyclophosphamide) Chemotherapy With G-CSF (Granulocyte Colony-Stimulating Factor) Followed by Infusional Taxol (Paclitaxel) as Adjuvant Treatment for High Risk Stage II and Stage III Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940145; 94-C-0145
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: 14-Day Cycle; Dose Intensity; Filgrastim; Lymph Node Positive; Non-Cross Resistant
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Granulocyte Colony-Stimulating Factor; Paclitaxel

INTERVENTIONS:
Drug: Adriamycin
Drug: cyclophosphamide
Drug: G-CSF
Drug: paclitaxel

SUMMARY:
This is a pilot feasibility trial of AC (Adriamycin, cyclophosphamide) chemotherapy with G-CSF (filgrastim) followed by infusional Taxol (paclitaxel) as adjuvant treatment for patients with high risk stage II and stage III breast cancer. Cycles will be 14 days in duration. After 3 fourteen day cycles of AC with filgrastim, patients will be treated with 3 fourteen day cycles of 96 hour infusional paclitaxel. The goal of this study will be to assess the toxicity and feasibility of administering dose-intensive AC chemotherapy followed by infusional paclitaxel in 14 day cycles.

DETAILED DESCRIPTION:
This is a pilot feasibility trial of AC (Adriamycin® (Registered Trademark), cyclophosphamide) chemotherapy with G-CSF (filgrastim) followed by infusional Taxol® (Registered Trademark) (paclitaxel) as adjuvant treatment for patients with high risk stage II and stage III breast cancer. Cycles will be 14 days in duration. After 3 fourteen day cycles of AC with filgrastim, patients will be treated with 3 fourteen day cycles of 96 hour infusional paclitaxel. The goal of this study will be to assess the toxicity and feasibility of administering dose-intensive AC chemotherapy followed by infusional paclitaxel in 14 day cycles.

ELIGIBILITY:
Recently diagnosed patients with histologically proven Stage II breast cancer who have 4 or more positive lymph nodes or patients with stage III breast cancer are eligible for this study.

Patients will be eligible for study either before or after receiving adjuvant radiation therapy.

Patients with stage III disease will be eligible to receive this regimen as neo-adjuvant chemotherapy or as adjuvant therapy if surgery was performed prior to patient referral.

Patients must be previously untreated with chemotherapy.

There must be no history of previous malignancy except for cured non-melanoma skin cancer (basal or squamous cell carcinoma), cervical cancer in situ, or a past malignancy that has been inactive for over 5 years. Patients with a prior history of lower stage contralateral breast cancer, treated with surgery, and/or radiation, but not chemotherapy, are eligible for this study.

Performance status (Karnofsky scale) must be greater than 70; ECOG 0 to 2.

Absolute granulocyte count greater than 1500 per microliter and platelet count greater than 100,000 per mm(3).

Liver function tests (SGOT, and total bilirubin) should be less than 2X upper limits of normal. Serum creatinine should be less than 1.7 or creatinine clearance should be greater than 45 ml per min.

The patient must be able to give an informed consent, and to return to NCI for treatment and adequate follow-up for the period the protocol requires.

Patients must be greater than or equal to 18 years of age.

Patients and/or their partners must be willing to practice a non-hormonal method of contraception during therapy and for 6 months following therapy.

Patients who are poor medical or psychiatric risks because of nonmalignant systemic disease which would preclude them from being subjected to any treatments in this protocol are excluded.

Patients must have a normal ejection fraction by MUGA scan and have no angina. Patients should not currently require therapy for cardiac arrhythmias, congestive heart failure, or coronary artery disease.

No patients with a history of symptomatic CNS disease.

No patients with allergy to any study medication.

No pregnant or lactating women.

Patients with bleeding disorders are ineligible for study entry as are patients requiring chronic anticoagulation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 1994-05; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Jones RB, Holland JF, Bhardwaj S, Norton L, Wilfinger C, Strashun A. A phase I-II study of intensive-dose adriamycin for advanced breast cancer. J Clin Oncol. 1987 Feb;5(2):172-7. doi: 10.1200/JCO.1987.5.2.172. PMID 3806165
- [Background] Wheeler RH, Ensminger WD, Thrall JH, Anderson JL. High-dose doxorubicin: an exploration of the dose-response curve in human neoplasia. Cancer Treat Rep. 1982 Mar;66(3):493-8. PMID 7060037
- [Background] Hryniuk W, Bush H. The importance of dose intensity in chemotherapy of metastatic breast cancer. J Clin Oncol. 1984 Nov;2(11):1281-8. doi: 10.1200/JCO.1984.2.11.1281. No abstract available. PMID 6387060